CLINICAL TRIAL: NCT01647269
Title: A Randomised, Controlled, Crossover Trial of Bilateral Deep Brain Stimulation to the Globus Pallidus Internum in Severe Tourette Syndrome
Brief Title: A Trial of Bilateral Deep Brain Stimulation to the Globus Pallidus Internum in Tourette Syndrome
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University College, London (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: UCL 11/0226
Record Dates: First submitted 2012-07-16; First posted 2012-07-23 (Estimated); Last update posted 2015-03-19 (Estimated); Status verified 2015-03

CONDITIONS: Tourette Syndrome
MeSH Terms: conditions — Tourette Syndrome

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- DBS Off first (Experimental)
  Interventions: Procedure: Bilateral GPi Deep Brain Stimulation
- DBS On First (Experimental)
  Interventions: Procedure: Bilateral GPi Deep Brain Stimulation

INTERVENTIONS:
Procedure: Bilateral GPi Deep Brain Stimulation — Bilateral GPi Deep Brain Stimulation

SUMMARY:
The purpose of this study is to investigate whether deep brain stimulation (DBS) of the globus pallidus internum (GPi) can alleviate tics in Gilles de la Tourette syndrome (GTS) and whether this treatment has any influence on social, psychological and behavioral disability and quality of life.

DETAILED DESCRIPTION:
This study is aimed at adults who have severe Tourette syndrome and who have found that conventional treatments, such as drugs, do not control their symptoms sufficiently or cannot be tolerated.

The first two clinic visits will involve assessments. Participants will fill in a number of questionnaires and be examined by a psychiatrist and a neurologist. At the second visit, the patient will provide consent for participation and will undergo formal tests to find out if the participant is suitable and willing to undergo the research study and to record the type and severity of their Tourette syndrome symptoms.

The third visit will be an admission to hospital to have the deep brain stimulation (DBS) devices implanted. The admission to hospital should be around five days in duration.

At the first post operative follow-up visit, the patient will be placed into a "stimulator on" group or a "stimulator off" group. To try and make sure that these groups are the same to start with, each patient is put into a group by chance (randomly). This visit will take place around six weeks after surgery. In this trial, the participant will have an equal chance of being in the "on" or the "off" group first. This trial is also a "blinded" trial, neither the patient nor the researchers performing the assessments will know which group the patient is in.

At the next visit, 3 months later, the patient will have a further assessment. If their stimulators have been "on" for the first 3 months, they will be switched off. If they have been "off" they will be switched on.

At the next visit, 3 months later, the patient will be assessed again and then given the opportunity to carry on the trial with the stimulators switched on for long term follow up.

ELIGIBILITY:
Inclusion Criteria:

1. The participant must be adult with stable Tourette syndrome.
2. The participant must have a chronic and severe tic disorder with severe functional impairment, with a Yale Tourette Severity Scale score of at least 35/55 for at least 12 months prior to surgery.
3. The participant must have failed conventional medical treatment at therapeutic doses of three classes of medication.
4. The participant must not be suitable for behavioural intervention or that this intervention is inappropriate or unsuccessful.
5. The participant must have been on stable and optimised treatment of co-morbid conditions for at least 6 months.
6. The participant must be actively involved with and compliant with any psychosocial interventions.
7. The patient must be compliant with treatment plans.

Exclusion Criteria:

1. The tic disorder is attributable to any other condition.
2. Any other medical or psychiatric disorders that substantially increase the risk of a failed procedure or that would significantly impede recovery.
3. Psychosocial factors which might impede operative and post-operative care and research participation.
4. Coagulation problems
5. Other disease compromising life expectancy
6. Patient likely to benefit from psychological intervention
7. Patient unwilling to co-operate with post operative assessment and care
8. Pregnancy.
9. Participant under 20 years old.

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2011-07; Primary Completion 2014-11 (Actual); Study Completion 2014-11 (Actual)

PRIMARY OUTCOMES:
Change in Yale Global Tic Severity Scale | Three months after stimulation switched ON v three months after stimulation switched OFF
  The Change in Scores on the Yale Global Tic Severity Scale will be compared between defined periods with stimulation switched ON v stimulation switched OFF.

SECONDARY OUTCOMES:
Change in Modified Rush Video Rating scale | Three months after stimulation switched ON v three months after stimulation switched OFF
Change in Yale Brown Obsessive Compulsive Scale | Three months after stimulation switched ON v three months after stimulation switched OFF
Change in Neuropsychiatric Inventory | Three months after stimulation switched ON v three months after stimulation switched OFF
Change in Tourette Quality of life scale | Three months after stimulation switched ON v three months after stimulation switched OFF
Change in MOVES scale | Three months after stimulation switched ON v three months after stimulation switched OFF
Change in Beck Depression Inventory | Three months after stimulation switched ON v three months after stimulation switched OFF

CONTACTS AND LOCATIONS:
Overall Officials: Thomas Foltynie, MBBS PhD, Principal Investigator — UCL Institute of Neurology
Locations (1):
- UCL Institute of Neurology, London, United Kingdom

REFERENCES:
- [Derived] Kefalopoulou Z, Zrinzo L, Jahanshahi M, Candelario J, Milabo C, Beigi M, Akram H, Hyam J, Clayton J, Kass-Iliyya L, Silverdale M, Evans J, Limousin P, Hariz M, Joyce E, Foltynie T. Bilateral globus pallidus stimulation for severe Tourette's syndrome: a double-blind, randomised crossover trial. Lancet Neurol. 2015 Jun;14(6):595-605. doi: 10.1016/S1474-4422(15)00008-3. Epub 2015 Apr 14. PMID 25882029